CLINICAL TRIAL: NCT00744614
Title: Use Of Capnography As Surrogate Measure Of PC02 In Medical ICU Patients
Brief Title: Use Of Capnography As Surrogate Measure Of PC02 In Medical Intensive Care Unit (ICU) Patients
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator (central contact) has left the organization and requests the study be terminated
Sponsor: Lahey Clinic (Other)
Responsible Party: David Riker, M.D., Lahey Clinic, Inc.
Other Study IDs: 2007-115
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: PC02; Respiratory Rate; Arterial blood gas; Intubation; Capnography
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Medical Intensive care unit patients with asthma, COPD, ILD or coronary disease who are at risk of intubation
  Interventions: Procedure: Capnography

INTERVENTIONS:
Procedure: Capnography — A technique for monitoring the concentration or partial pressure of CO2 levels in respiratory gases

SUMMARY:
The purpose of this study is to evaluate the use of Capnography (Continuous recording of the carbon dioxide content of expired air)as an alternative test to measure PC02 levels in patients with asthma, chronic obstructive pulmonary (COPD,interstitial lung disease(ILD)or coronary disease who are at risk of intubation.

DETAILED DESCRIPTION:
This is a prospective study to evaluate the usefulness of capnography as a non-invasive, accurate method of measuring of PC02 levels in medical intensive care unit patients with asthma, COPD, ILD, or coronary disease who are at risk of intubation.

ELIGIBILITY:
Inclusion Criteria:

* Medical Intensive Care Patients
* Not intubated
* Age 18 or older
* History of any one of the following: asthma, COPD, ILD, or coronary disease

Exclusion Criteria:

* Sepsis
* Life expectancy less than 1 month
* Requiring BIPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MICU patients who are at risk of intubation and who have a history of asthma, COPD, ILD or coronary disease.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
PCO2 level | 6 months

SECONDARY OUTCOMES:
Time to intubation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David R. Riker, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Torok SS, Leuppi JD, Baty F, Tamm M, Chhajed PN. Combined oximetry-cutaneous capnography in patients assessed for long-term oxygen therapy. Chest. 2008 Jun;133(6):1421-1425. doi: 10.1378/chest.07-0960. Epub 2008 Mar 13. PMID 18339783